CLINICAL TRIAL: NCT06026267
Title: Efficacy of Conventional Dose Protocol vs Low Dose Protocol Albumin Use in Patients With Cirrhosis and High Risk Spontaneous Bacterial Peritonitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-59
Record Dates: First submitted 2023-08-17; First posted 2023-09-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Liver Cirrhosis; Spontaneous Bacterial Peritonitis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose Arm+Standard Medical therapy (Active Comparator): Human Albumin 20% 1.5 g/kg body weight (Maximum 100g) on day 1 after the diagnosis, followed by 1 g/kg body weight (Maximum 100g)on day 3 along with standard medical therapy.
  Interventions: Biological: 20% High Dose Albumin; Other: Standard Medical Treatment
- Reduced Dose Albumin+Standard Medical therapy (Experimental): Human Albumin 20% 1.0 g/kg body weight (Maximum 100g) on day 1 after the diagnosis, followed by 0.5 g/kg bodyweight (Maximum 100g) on day 3 along with standard medical therapy.
  Interventions: Other: Standard Medical Treatment; Biological: 20% Reduced Dose Albumin

INTERVENTIONS:
Biological: 20% High Dose Albumin — A]. Patients in the conventional albumin Arm will receive Human Albumin 20% 1.5 g/kg body weight (Maximum 100g) on day 1 after the diagnosis, followed by 1 g/kg bodyweight (Maximum 100g)on day 3 along with standard medical therapy.
  Duration of albumin over 24 hours.
  Arms: High Dose Arm+Standard Medical therapy
Other: Standard Medical Treatment — Standard Medical Treatment
Biological: 20% Reduced Dose Albumin — B]. Patients in the low dose albumin Arm will receive Human Albumin 20% 1.0 g/kg body weight (Maximum 100g) on day 1 after the diagnosis, followed by 0.5 g/kg bodyweight (Maximum 100g) on day 3 along with standard medical therapy.
  Duration of albumin over 24 hours.
  Arms: Reduced Dose Albumin+Standard Medical therapy

SUMMARY:
The role of Albumin in prevention and Treatment of Acute Kidney Injury (AKI) in patients with Spontaneous Bacterial Peritonitis (SBP) who are at high risk of AKI development has been clearly defined, which decreases the morbidity and mortality. However the conventional dose recommended by the guidelines is usually not tolerated by the Indian population. Investigator propose that the low dose is as beneficial as the standard dose in patients with high risk SBP in the prevention/progression of renal dysfunction in cirrhotic patients with high risk spontaneous bacterial peritonitis. If confirmed, these results could support a significant cost reduction in the management of ascites in cirrhotic patients and decrease the side effects of the volume overload in the patient of the cirrhosis.

DETAILED DESCRIPTION:
Hypothesis Alternate Hypothesis: Low dose albumin is as effective as conventional dose albumin in cirrhosis with high risk SBP patients having AKI development or progression by day 4.

Aim:-To compare the efficacy and safety of low dose albumin with conventional dose albumin in AKI development or progression in patients with cirrhosis and high risk spontaneous bacterial peritonitis.

Study population: Patients of age > 18 years of age with cirrhosis of liver who are admitted in ward/ICU diagnosed with high risk SBP.

Study design: Randomized controlled trial Study period:1.5year Sample size: 300 (150 cases in each group) Assuming that the rate of AKI development in conventional dose albumin group - 10% and low dose albumin group 15%, Power- 80%, Alpha- 10% ONE SIDED, Non inferiority limit- 5, cases needed to enroll are 270, further assuming 10% dropout, investigator decided to enroll total 300 cases, randomly allocated with 150 cases in each arm by block randomization method with Block size of 10 Cases will be randomly allocated in 2 groups by block randomization method with block size taken as 10.

STATISTICAL ANALYSIS:

Continuous variables- Mean +/- SD Categorical variables as percentages (%) or Frequencies Student t test will be applied in continuous data compared with two groups Survival analysis like Cox-Regression model and Kaplan-Meir plots will be plotted to find the possible factors responsible for mortality Besides these, Intent to treat (ITT) and Per Protocol (PP) will be done at the time of data analysis.

Adverse effects:

Patients receiving Albumin may experience Nausea, Vomiting, Fever with chills, dyspnea Wheezing, Volume overload, Anaphylactic reaction

Stopping rule of study:

Adverse reaction to drug Cardiopulmonary compromise

ELIGIBILITY:
Inclusion Criteria:

1. Age >18years
2. Cirrhosis with SBP (community acquired /Health care associated/ nosocomial)
3. High risk SBP : Patients with S Bil >4 mg/dL and/or s creat > 1 mg/dl at presentation

Exclusion Criteria:

1. Antibiotic treatment within one week before the diagnosis of SBP (except for prophylactic treatment with norfloxacin)
2. Significant cardiac failure, pulmonary disease
3. Known CKD or findings suggestive of organic nephropathy (proteinuria, haematuria, or abnormal findings on renal USG)
4. Hepatocellular carcinoma
5. HIV infection
6. GI bleed within 1 month before the study
7. Grade 3 to 4 hepatic encephalopathy
8. Shock (MAP < 65)
9. Serum creatinine level of > 3 mg/decilitre
10. Presence of any potential causes of dehydration (such as diarrhea or an intense response to diuretic treatment within one week before the diagnosis of SBP).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients developing new AKI or having progression of AKI by day 4. | Day 4

SECONDARY OUTCOMES:
Resolution of Spontaneous Bacterial Peritonitis by day 5 | Day 5
  Resolution is defined as decrease in ascitic fluid PMN > 25% from baseline
Change on Serum Ascites Albumin Gradient (SAAG) in both the groups. | Day 5
Change in cell count (PMN) in both groups. | Day 5
Changes in PRA levels from baseline to day 7 | day 7
Changes in TNF-alpha levels from baseline to day 7 | day 7
Changes in IL-6 levels from baseline to day 7 | day 7
Changes in endotoxin levels from baseline to day 7 | day 7
Changes in renal resistive index from baseline to day 7 | day 7
Number of patients with development of complications in both groups | 90 days
Number of Participants with changes in ProBNP from baseline to day 4 or if shortness of breath occurs | Day 4
Number of Participants with changes in vWF-Ag from baseline to day 4 | Day 4
Number of patients expired in both the groups | Day 7
Number of patients expired in both the groups | Day 28
Number of patients expired in both the groups | Day 90
Duration of hospital stay | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided